CLINICAL TRIAL: NCT04798105
Title: Modulation of Probabilistic Selection Task Performance Based on Anodal tDCS of dlPFC, Eye Blink Rate, Extraversion and Impulsiveness
Brief Title: Predictors of Probabilistic Selection Task Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles Darwin University (Other)
Responsible Party: Principal Investigator, Luca Aquili, Lecturer (B) in Psychology, Charles Darwin University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CDULA2021
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Learning; Lack of (Specific)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS sham (Sham Comparator): Transcranial direct current stimulation (tDCS) of the dorsolateral prefrontal cortex (dlPFC) in sham mode.
  Interventions: Behavioral: Effects of tDCS of dlPFC on Probabilistic Selection Task
- tDCS anodal (Active Comparator): Transcranial direct current stimulation (tDCS) of the dorsolateral prefrontal cortex (dlPFC) in anodal/excitatory mode.
  Interventions: Behavioral: Effects of tDCS of dlPFC on Probabilistic Selection Task

INTERVENTIONS:
Behavioral: Effects of tDCS of dlPFC on Probabilistic Selection Task — Predictors of Probabilistic Selection Task Performance including anodal tDCS of dlPFC, eye blink rate, extraversion and impulsiveness

SUMMARY:
The project aims to investigate whether tDCS has an effect on reward and punishment learning sensitivity. Further, whether tDCS will modulate extraversion and impulsivity personality traits, and eye-blink-rate's effect on learning. For instance, trait extroversion in past research is linked to the dopamine neurotransmitter system, where it is thought that extreme low and high levels are detrimental to cognitive performance. Since tDCS has been shown to increase dopamine levels, it is thought that people who are already high in dopamine may experience less benefit (or even impairment) on cognitive performance following tDCS.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of a non-invasive, low intensity and risk, brain stimulation technique known as transcranial direct current stimulation (tDCS) on the way people learn in a computer administered cognitive task. This will be achieved by comparing participants' performance on this task after receiving placebo 'sham' tDCS in one experimental session, and real 'treatment' tDCS in another experimental session. Neither the researcher administering the session or the participant will be aware of which form of tDCS is being used. Previous research indicates that tDCS of the left dorsolateral prefrontal cortex brain region stimulates the release of a chemical neurotransmitter, dopamine, that is linked to reward and punishment processing, and implicated in conditions such as addiction and Parkinson's disease.

The computerized cognitive learning task presents participants with pairs of six different symbols and asks them to choose one of these. In the first half of the task, participants receive visual feedback (correct or incorrect; +$0.10 or -$0.10) and the symbols are preprogrammed to be rewarded or punished for. In the second part of the task, participants are tested on the same task but do not receive feedback.

Further, the effect of participants' personality characteristics (specifically extraversion and impulsivity), as well as eye-blink-rate, on cognitive learning performance will be investigated, as this is known to be influenced by tDCS. Past research suggests that people may respond differently to tDCS based on individual differences in these personality traits, that are linked at a brain circuits level. Participants will be assessed on extraversion and impulsivity personality traits using pen and paper, self-report questionnaires. Similarly, eye-blink-rate is linked to the aforementioned brain neurotransmitter, dopamine, and will be assessed by manually counting of blinks in a video recording of the participant focusing on a stationary point.

ELIGIBILITY:
Inclusion Criteria:

* Either male or female
* You are aged between 18 and 50 years
* You are in good health
* You agree to fast 3 hours prior to testing

Exclusion Criteria:

* Suffer from cardiac, hepatic, renal, and/or neurological disorders
* Have damaged or diseased skin on your face and scalp, or a sensitive scalp
* Have a history of alcohol or drug addiction, or severe psychiatric illness
* Are receiving drug treatment which may lower seizure threshold (i.e. epilepsy)
* Are pregnant
* Are sleep deprived (less than 6 hours a day)
* Have metallic dental fillings, orthodontic appliances, a cardiac pacemaker, cochlear implant, and/or surgical clips
* Have a history of migraine or headaches

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-10-22 (Estimated); Study Completion 2021-10-22 (Estimated)

PRIMARY OUTCOMES:
Change in Probabilistic Selection Task (PST) performance from pre tDCS to post tDCS | PST is tested prior to tDCS administration at time 0 (baseline) and following tDCS (approximately 50 minutes into the experiment) for both tDCS sham and tDCS anodal
  Accuracy (%) and reaction times on the above task

CONTACTS AND LOCATIONS:
Locations (1):
- Charles Darwin University, College of Health & Human Sciences, Darwin, Northern Territory, Australia

IPD SHARING:
Plan to Share IPD: No